CLINICAL TRIAL: NCT03288025
Title: Pulmonary Arterial Hypertension Improvement With Nutrition and Exercise (PHINE) A Randomized Controlled Trial
Brief Title: Pulmonary Arterial Hypertension Improvement With Nutrition and Exercise (PHINE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gustavo A Heresi, MD, MS, Staff, Pulmonary Medicine, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-260; R01HL130209 (NIH)
Record Dates: First submitted 2017-08-31; First posted 2017-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension; Insulin Resistance
Keywords: Insulin Resistance; Inflammation; Right Ventricular Function; Metabolism; Glucose
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Insulin Resistance; Inflammation | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrition and Exercise (Experimental): 5 days a week of moderate exercise and biweekly diet counseling on Low Glycemic Index/ Mediterranean Diet for 12 weeks.
  Interventions: Behavioral: Nutrition and Exercise
- Standard of Care (No Intervention): Counseling at baseline on diet as recommended by USDA and on the benefits of regular aerobic exercise.

INTERVENTIONS:
Behavioral: Nutrition and Exercise — 5 times a week exercise training and biweekly diet counseling for 12 weeks.
  Arms: Nutrition and Exercise

SUMMARY:
The purpose of this study is to investigate the extent to which diet and exercise may improve PAH through the modulation of insulin sensitivity. The central hypothesis is that dysregulated glucose metabolism elicits a response in PAH patients that can be modified by exercise and diet, thereby leading to improvements in pulmonary vascular disease.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) leads to premature death as a consequence of increased pulmonary vascular resistance and right heart failure. PAH-targeted therapies developed over the past 20 years target excessive vasoconstriction. However, the pathobiology of PAH is more complicated, and includes dysregulated vascular cell proliferation, cellular metabolic abnormalities, and inflammation. Even with modern PAH therapies, current outcomes remain poor, with an estimated 3-year survival rate of only 55%. Thus, there is a clear need for more effective therapies, based on better understanding of the pathobiology of the disease.

Insulin resistance has emerged as a potential new mechanism in PAH. Animal models of insulin resistance are associated with PAH, which reverses with the administration of insulin sensitizing drugs. Over the past decade there has been an epidemiologic shift in PAH, where the disease is increasingly observed in older, obese, and diabetic subjects. Low levels of high-density lipoprotein cholesterol in PAH, a feature of insulin resistance, have been observed and found to be a strong independent predictor of PAH mortality. Elevated glycosylated hemoglobin (HbA1c) also correlates with PAH diagnosis and severity. As measured by the OGTT, idiopathic PAH patients have not only insulin resistance, but also an inability to mount an appropriate insulin response to a glucose challenge. These data point to dysfunction in the pancreatic beta cells of PAH patients. It is known that an exercise and low glycemic index diet intervention improves insulin sensitivity in pre-diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18-75 years old
* Group 1 PAH, including idiopathic, heritable, drugs and toxin induced, and PAH associated with connective tissue disease, HIV infection and congenital heart disease
* NYHA Class II or III
* ≥ 1 PAH-targeted therapy with a stable dose for ≥ 2 months
* Stable dose of diuretics and rate of supplemental oxygen for the preceding 2 months

Exclusion Criteria:

* Decompensated Right Heart Failure
* NYHA Class IV
* Syncope within the previous 3 months
* Cardiac Arrhythmia (except for controlled atrial fibrillation or flutter)
* Baseline supplemental O2 > 4 LPM
* Portal Hypertension
* Pulmonary hypertension due to Lung Disease and Hypoxia
* Pulmonary Hypertension due to Left Heart Disease
* Chronic Thromboembolic Pulmonary Hypertension
* Pulmonary Hypertension associated with systemic diseases such as hematological disorders and sarcoidosis
* Type 2 Diabetes
* Evidence of cardiac ischemia on a graded exercise test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | 5 years
  Assessed by the frequently-sampled intravenous glucose tolerance test. Units of assessment in min/uU*mL

SECONDARY OUTCOMES:
Right Ventricular Global Peak Longitudinal Strain | 5 years
  Assessed by the Doppler Echocardiography 2D longitudinal speckle tracking. Units of assessment in percent.

CONTACTS AND LOCATIONS:
Overall Officials: Raed Dweik, MD, Principal Investigator — The Cleveland Clinic; Gustavo Heresi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No